CLINICAL TRIAL: NCT01364948
Title: Effect of Topical Oil Application on Trans-epidermal Water Loss (TEWL) in Preterm Very Low Birth Weight (VLBW) Infants - A Randomized Clinical Trial
Brief Title: Effect of Coconut Oil Application in Reducing Water Loss From Skin of Premature Babies in First Week of Life (TEWL)
Acronym: TopOilTewl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr Sushma Nangia, Division of Neonatology, Department of Pediatrics, AIIMS, New Delhi, India
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A-28/Dec 2005
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2005-12

CONDITIONS: Trans Epidermal Water Loss (TEWL)
Keywords: Preterm; VLBW; Coconut Oil application; Trans epidermal water loss; Weight gain
MeSH Terms: conditions — Premature Birth; Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coconut oil application (Experimental): The oil (coconut oil) was applied by the trained nurse to the entire body surface of infant except the face two times a day starting at 12 hrs of life. Four ml of coconut oil was applied using both hands of the caregiver in four strokes. First stroke was from the clavicles over the chest and abdomen till the groin, second from the front of thighs over the knee and leg upto the sole, the third one from the shoulders over the arm and forearm till the palm continuing medially over the forearm and arm till the axilla and the final stroke was used for the back, starting from the upper back, continuing over the back of the thighs till the heel. Just prior to the first application, and thereafter prior to the subsequent applications the TEWL was recorded using the portable closed chamber evaporimeter. The oil application was continued twice daily (every 12 hrs at the same time as the hour of birth e.g. 11 am and 11pm) till the completion of the seventh day (168 hrs of life).
  Interventions: Other: Coconut oil application
- No Oil Application (No Intervention): Babies in this group were not subjected to oil application. TEWL measurement was recorded every 12 hrs for the first week of life, at the same time as the hour of birth.
  Interventions: Other: No oil application

INTERVENTIONS:
Other: Coconut oil application — Four ml coconut oil application twice daily for first week
  Arms: Coconut oil application
Other: No oil application — Oil application was not done
  Arms: No Oil Application

SUMMARY:
The skin of newborn infants is immature and ineffective as a barrier. Preterm skin exhibits even more vulnerability to the environment due to poor self regulatory heat mechanisms, paucity of fatty tissue and its thinness. Most preterm babies lose up to 13% of their weight as water loss from their skin during the first week of life. Many strategies have been utilized by neonatologists to decrease this water loss. Oil application on the skin can act as a non permeable barrier and can help in reducing water loss from the skin. Edible coconut oil, often used for traditional massage of babies by Indian communities, is culturally acceptable and Hence the investigators decided to undertake this study to objectively assess the reduction in water loss from skin after oil application

ELIGIBILITY:
Inclusion Criteria:

All preterm babies born at the study center with birth weight < 1500gms were eligible for inclusion in the study.

Exclusion Criteria:

1. Babies with birth weight less than 750 gms at birth
2. Babies with major congenital malformations.
3. Babies with severe asphyxia, hydrops and shock.
4. Babies with congenital diseases of skin associated with skin breach or denudation of skin precluding oil application
5. Babies with preexisting skin infection such as multiple furuncles (2 or more skin areas - each limb, head, chest, abdomen and back are the individual areas that will be taken as one area

Ages: 12 Hours to 168 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Trans Epidermal Water Loss(TEWL) | first 7 days of life
  TEWL was measured using evaporimeter(Vapometer, Delfin Technologies limited, Kuopio, Finland) at 12 hours of age and thereafter every 12 hours during the first week of life (168 hrs of life)

SECONDARY OUTCOMES:
Weight | Weight first 7 days of life and 40 weeks postmenstrual age
  The weight of the neonate was recorded at birth and daily during the first week of life. The weight in grams and weight gain in grams/kilogram/day was measured at 40 weeks post conceptional age.
Skin condition Score | Skin condition Score at day 7 of life
  Skin Condition Score was measured using 'Lane and Drost' Score.This score has 9 scores from 1 to 9, 1 depicting the best skin state and 9 the worst with erythema, blistering & oozing over the entire area.
Skin colonization pattern | Skin colonization pattern at day 7 of life
  The skin swab cultures were sent after 1week of life to assess for skin colonization

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sushma Nangia, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi, India